CLINICAL TRIAL: NCT05160883
Title: Neuroimaging Changes in Hereditary Ataxia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Wulab-MRI in HA
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Ataxia
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to investigate the neuroimaging changes of hereditary ataxia patients, especially in the SCA3 patients in preclinical or mild stage.

ELIGIBILITY:
Inclusion Criteria:

* genetically diagnosed as Spinocerebellar ataxia

Exclusion Criteria:

* deny to follow-up

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with hereditary ataxia
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
neuroimaging information | from 2021 to 2025
  neuroimaging information approached by MRI, including 3D-T1, T2, DTI, rsfMRI, SWI, ASL were collected

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China